CLINICAL TRIAL: NCT01349452
Title: Ganciclovir 0,15% Ophthalmic Gel in the Treatment of Adenovirus Keratoconjuntivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Simone Tiemi Yabiku, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAN2011
Record Dates: First submitted 2011-04-29; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-04

CONDITIONS: Conjunctivitis, Viral; Adenoviridae Infections
Keywords: Conjunctivitis, Viral; Adenoviridae Infections; Ganciclovir; Adenovirus Keratoconjunctivitis; Treatment of viral conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Viral; Adenoviridae Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ganciclovir (Experimental)
  Interventions: Drug: Ganciclovir
- Artificial tear (Sham Comparator)
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Drug: Ganciclovir — Ganciclovir 0.15% Ophthalmic gel
  Arms: Ganciclovir
Drug: Artificial tear — Artificial tear 5 times per day
  Arms: Artificial tear

SUMMARY:
Ganciclovir ophthalmic gel delivers multiple advantages in the treatment and prophylaxis of herpetic keratitis and shows potential for effectiveness against other viral ocular infections. The majority of adenoviral conjunctivitis will resolve without damaging vision, however, the investigators have no way to determine which cases will progress to ocular complications such as corneal infiltrates and pseudomembranes. Our purpose is to evaluate the efficacy of the Ganciclovir gel 0.15% in preventing ocular complications after adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* onset of symptoms for five days or less
* eighteen years old or more
* not pregnant or breastfeeding
* be able to understand and sign the consent term

Exclusion Criteria:

* use of antibiotic or corticoid 30 days before
* monocular vision
* keratopathy or other ocular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
improvement of symptoms of conjunctivitis (pain relief) | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Simone T Yabiku, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Yabiku ST, Yabiku MM, Bottos KM, Araujo AL, Freitas Dd, Belfort R Jr. [Ganciclovir 0.15% ophthalmic gel in the treatment of adenovirus keratoconjunctivitis]. Arq Bras Oftalmol. 2011 Nov-Dec;74(6):417-21. doi: 10.1590/s0004-27492011000600007. Portuguese. PMID 22331114